CLINICAL TRIAL: NCT07319442
Title: Long-term Observation of IBD Patients, a Nationwide German IBD Registry "CEDUR"
Brief Title: CEDUR - German IBD Registry
Acronym: CEDUR
Status: Recruiting | Type: Observational
Sponsor: ImmunoRegister gUG (Other)
Responsible Party: Sponsor
Other Study IDs: HW-PV5539
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis (UC); Indeterminate Colitis; Crohn Disease (CD)
Keywords: IBD; Registry; Crohn's disease; Ulcerative Colitis; Real-world-data; Germany; Quality of care; pharmaeconomics; safety; long-term follow-up; patient journey; treatment algorithm
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CEDUR registry systematically collects real-world data on inflammatory bowel disease (IBD) patients in Germany. The registry aims to assess quality of care, disease activity, treatment effectiveness, safety, and pharmacoeconomic aspects under routine clinical conditions.

DETAILED DESCRIPTION:
CEDUR is a multicenter, web-based, observational registry for adult IBD patients in Germany. The registry includes Crohn's disease, ulcerative colitis, and indeterminate colitis. Data are collected prospectively from physicians and patients, covering clinical parameters, quality of life, treatment patterns, and safety outcomes. The registry supports the evaluation of care quality, cost-effectiveness, and long-term therapy outcomes under real-life conditions.

ELIGIBILITY:
Inclusion Criteria:

* Crohn Disease Ulcerative Colitis Indterminate Colitis

Exclusion Criteria:

* Other gastrointestinal disorders than above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with a confirmed diagnosis of Crohn's disease, ulcerative colitis, or indeterminate colitis who receive routine medical care in Germany. Patients are recruited by participating gastroenterologists in hospitals and private practices and are followed prospectively within the CEDUR registry for long-term observation of disease course, treatment patterns, safety, and quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2036-05 (Estimated); Study Completion 2036-05 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) | Up to 10 years of follow-up
  The Crohn's Disease Activity Index (CDAI) is a composite clinical score assessing disease activity in patients with Crohn's disease. It incorporates eight variables including stool frequency, abdominal pain, general well-being, extraintestinal manifestations, and laboratory parameters. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity.
Partial Mayo Score | Up to 10 years of follow-up
  The Partial Mayo Score is a clinical index used to assess disease activity in ulcerative colitis. It includes stool frequency, rectal bleeding, and physician's global assessment, with scores ranging from 0 to 9. Higher scores indicate more severe disease activity.
Mayo Score (Full Mayo Score) | Up to 10 years of follow-up
  The Mayo Score is a composite index used to assess disease activity in ulcerative colitis. It consists of four components: stool frequency, rectal bleeding, physician's global assessment, and endoscopic findings. Total scores range from 0 to 12, with higher scores indicating more severe disease activity.
Simple Endoscopic Score for Crohn's Disease (SES-CD) | Up to 10 years of follow-up
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) is an endoscopic index used to quantify mucosal disease activity in Crohn's disease. It assesses ulcer size, ulcerated surface, affected surface, and presence of strictures across bowel segments. Higher scores indicate more severe endoscopic disease activity.
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Up to 10 years of follow-up
  The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a validated patient-reported outcome measure assessing health-related quality of life in patients with inflammatory bowel disease. It consists of 10 items covering bowel, systemic, emotional, and social domains. Total scores range from 10 to 70, with higher scores indicating better quality of life.
PROMIS-10 Global Health Score | Up to 10 years of follow-up
  The PROMIS-10 Global Health is a validated patient-reported outcome measure assessing global physical and mental health. It consists of 10 items generating physical and mental health summary scores standardized to a T-score metric. Higher scores indicate better self-reported health status.
Bowel Urgency Score | Up to 10 years of follow-up
  The Bowel Urgency Score is a patient-reported measure assessing the severity and frequency of urgency to defecate. The range is from 0-10. Higher scores indicate greater bowel urgency and symptom burden.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Up to 10 years of follow-up
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a validated patient-reported outcome measure assessing fatigue and its impact on daily functioning in patients with chronic illness. It consists of 13 items, with total scores ranging from 0 to 52. Higher scores indicate less fatigue and better functional status.

SECONDARY OUTCOMES:
Change in Disease activity over time | Up to 10 years of follow-up
  Effectiveness of inflammatory bowel disease therapies will be assessed by longitudinal changes in validated disease activity indices, including clinical, endoscopic, and patient-reported outcome measures, during registry follow-up.
Treatment persistence (drug persistence) | Up to 10 years of follow-up
  Treatment persistence is defined as the duration of continuous therapy from initiation to discontinuation or switch of treatment for any reason during registry follow-up.
Incidence of adverse events and serious adverse events | Up to 10 years of follow-up
  Safety will be assessed by the frequency, type, and severity of adverse events (AEs) and serious adverse events (SAEs) reported by participating physicians during registry follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Howaldt, MD, Principal Investigator — ImmunoRegister gUG
Locations (1):
- ImmunoRegister gUG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the registry collects pseudonymized patient information under strict data protection regulations (GDPR) in Germany. Data are available only in anonymized and aggregated form for approved scientific analyses conducted by the Scientific Advisory Committee.

REFERENCES:
- See also: Official website of the sponsor organization ImmunoRegister gUG. — https://www.immunoregister.de